CLINICAL TRIAL: NCT06456242
Title: Using Contingency Management to Promote Adherence to Smoking Cessation Treatment
Brief Title: Contingency Management to Promote Smoking Cessation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DA055779
Record Dates: First submitted 2024-06-04; First posted 2024-06-13 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MedCM plus CounsCM (Experimental): Mobile Contingency Management for counseling attendance and medication intake
  Interventions: Behavioral: CounsCM+MedCM (Health Rewards)

INTERVENTIONS:
Behavioral: CounsCM+MedCM (Health Rewards) — Small financial incentives for completing quitline calls (CounsCM) plus small financial incentives for taking varenicline (MedCM).

SUMMARY:
Many hospitals and outpatient clinics often refer people who smoke to quitlines and provide prescriptions for smoking cessation medications, but patients rarely fully engage in counseling or use their cessation medications. This is a single-arm, open-label pilot study to provide feasibility metrics for a text-based contingency management (CM) intervention to increase engagement in smoking cessation treatment. All participants (N=20) will be referred to a state quitline and will receive a prescription for medication plus 12 weeks of a text-based CM intervention to increase engagement in quitline calls and varenicline utilization. The engagement of participants in quitline counseling will be tracked for 6 weeks and medication utilization for 12 weeks post-enrollment. The investigators will use mixed-methods to collect implementation and acceptability data to inform changes to the text-based contingency management (CM) intervention.

DETAILED DESCRIPTION:
Novel approaches are needed to engage people who smoke in treatment in a way that increases their odds of quitting. Contingency management (CM) interventions provide financial incentives to participants contingent on objective evidence of behavior change and are effective in enhancing medication adherence and treatment engagement for numerous health conditions, including tobacco dependence treatment. Critical gaps, however, remain in our knowledge regarding how best to deploy CM.

The goal of this study is to evaluate the acceptability and feasibility of combined CM for engaging patients in smoking cessation treatment. Participants (N=20) will receive "CounsCM" for engaging in five quitline calls and "MedCM" for utilizing varenicline over twelve weeks. CM payments will be automated and dispensed on a daily basis using a reloadable debit card. The investigators will use surveys and structured interviews to understand strengths, weaknesses, and areas for improvement.

ELIGIBILITY:
Inclusion Criteria:

* Smoked in the past 30 days
* Smoke at least 1 cigarette per day when they smoke
* ≥ 18 years old
* Kansas resident
* Speak/read English
* Access to a mobile phone
* Mobile phone receives text messages
* No varenicline contraindications (no acute renal impairment)
* Insurance coverage for varenicline
* Have no significant co-morbidity (i.e., life-threatening illness, communication barriers or altered mental status)
* Cognitively able to participate
* Physically able to participate
* Not pregnant/breastfeeding

Exclusion Criteria:

* Medically ineligible for varenicline
* Patient on smoking cessation medication within 2 weeks of admission date
* Patient already talked to quitline in the past 2 weeks.
* Patients participating in other quit smoking program or research study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of quitline calls completed | Week 6
  Completion of the five quitline calls over 6 weeks of treatment according to Kansas quitline reports
Proportion of varenicline pills taken | Week 12
  Varenicline intake over 12 weeks of treatment according to the smart pill dispenser counting

SECONDARY OUTCOMES:
Proportion of patients adherent to varenicline | Week 3
  Adherence biochemically verified using saliva samples, 1.0 ng/ml as the cutoff to distinguish between participants adherent and adherent
Proportion of self-reported varenicline pills taken | Week 3
  Self-reported use of varenicline from a timeline followback questionnaire assessing varenicline pills taken in each of the past 3 days
Proportion of patients with biochemically verified smoking abstinence | Week 12
  Biochemically confirmed 7-day point prevalence abstinence using the anabasine criteria cutoff of ≤ 2 ng/ml
Proportion of patients with self-reported smoking abstinence | Week 12
  Past 7 days self-reported smoking abstinence

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States